CLINICAL TRIAL: NCT06102551
Title: A Retrospective Study of Factors Associated With Postoperative Recurrence of Incisional Hernia Repair in the Abdominal Wall
Brief Title: A Retrospective Analysis of Incisional Hernia Repair's Postoperative Recurrence
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhijun Bao, Director, Fudan University
Other Study IDs: HuadongHosptialHernia01
Record Dates: First submitted 2023-09-23; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Incisional Hernia; Recurrent Hernia
MeSH Terms: conditions — Incisional Hernia; Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The primary group
- The recurrent group
  Interventions: Behavioral: Recurrence after surgery

INTERVENTIONS:
Behavioral: Recurrence after surgery — Recurrence after repair was the main outcome
  Groups: The recurrent group

SUMMARY:
ABSTRACT Purpose：A retrospective study was conducted among patients with incisional hernia in our hospital to analyse the factors associated with postoperative recurrence of abdominal wall incisional hernia.

Methods：Patients with a diagnosis of incisional hernia obtained from our hospital's electronic medical record system were divided into primary incisional hernia group and recurrent incisional hernia group according to whether or not they had a recurrence after surgery. Baseline information on these patients was recorded and statistically analysed after our review.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria: diagnosis of incisional hernia of the abdominal wall and primary; surgical treatment for hernia repair at our hospital; all patients originating from outpatient clinics rather than emergency clinics; age of 18 to 80 years at the time of admission; and those with a well-established preoperative examination.

Exclusion Criteria:

* Exclusion criteria: severe organ dysfunction (ASA score of IV, V, VI); unconsciousness and poor cooperation with various preoperative examinations; correction of other types of abdominal hernia by perfect examination after admission; incomplete necessary information.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * Inclusion criteria: diagnosis of incisional hernia of the abdominal wall and primary; surgical treatment for hernia repair at our hospital; all patients originating from outpatient clinics rather than emergency clinics; age of 18 to 80 years at the time of admission; and those with a well-established preoperative examination.
  Exclusion Criteria:
  * Exclusion criteria: severe organ dysfunction (ASA score of IV, V, VI); unconsciousness and poor cooperation with various preoperative examinations; correction of other types of abdominal hernia by perfect examination after admission; incomplete necessary information.
Sampling Method: Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Recurrent | 2017.1-2023.8
  Recurrence after surgery repair

CONTACTS AND LOCATIONS:
Locations (1):
- YiMing Lin, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No